CLINICAL TRIAL: NCT06436287
Title: Handwriting Analysis in Movement Disorders.
Status: Not yet recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Aditya Murgai, Assistant Professor in Neurology, Western University, Canada
Other Study IDs: 123953
Record Dates: First submitted 2024-05-06; First posted 2024-05-31 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Movement Disorders
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Diagnosed with a movement disorder
- Control: Healthy controls

SUMMARY:
Movement disorders are a group of neurological conditions that cause problems with movement, either in the form of excessive, reduced, or slow movements. Some commonly known movement disorders include Parkinson disease, dystonia, ataxia, and Tourette syndrome. Multiple movement disorders have unique handwriting characteristics that can be measured using an inkless pen and a digitalized tablet. Handwriting is a complex skill that requires a combination of cognition, motor planning, and visuomotor integration. Handwriting deteriorates in patients with neurodegenerative diseases.

This study aims to discern variations in the kinematics (movement patterns) involved in handwriting between individuals with movement disorders and healthy controls. Participants will be invited to carry out a series of handwriting tasks. The pen motions will be captured using an inkless pen and a digitizing tablet linked to a laptop. The entire set of tasks is designed to be completed within 30 minutes. The data will then be collected, processed, and analyzed utilizing a handwriting analysis software.

DETAILED DESCRIPTION:
Background: Handwriting is a complex skill that requires a combination of cognition, motor planning, and visuomotor integration. Various brain structures including the cerebral cortex, basal ganglia, and cerebellum are involved in learning and performing handwriting. Many neurological disorders impact these brain structures in unique ways, leading to distinct effects on handwriting. Changes in handwriting performance are a prominent feature of Parkinson disease (PD), ataxias, and other movement disorders. Handwriting analysis can serve as a tool to distinguish and monitor the progression of movement disorders. Patients suffering from PD exhibit impairments of previously learned motor skills, including handwriting. It has been demonstrated that patients in the early stages of Parkinson disease exhibit variations in handwriting when compared to healthy individuals. The current research will investigate kinematics, visuospatial adaptation, and learning in different movement disorders through handwriting analysis.

Data collection and Measurement techniques: The subject will be seated comfortably at a table with the digitalized tablet positioned to allow a natural writing position for the subject. Pen movements will be recorded using a non-inking pen and Wacom Cintiq 16-inch digitizing tablet connected to a laptop. A practice session will be provided to each participant to familiarize them with the inkless writing pen and tablet. Before each task, participants will be given instructions on how to perform the task. Participants will be instructed to complete several writing exercises aimed at evaluating various aspects of their handwriting skills. Each task will be repeated multiple times and the entire set of handwriting exercises will be completed within 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

(1) Diagnosed with a movement disorder.

Exclusion Criteria:

1. Action tremor or weakness in the dominant hand interfering with writing task.
2. Unable to write or understand English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Movement disorder patients will be recruited from the London Movement Disorder Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Primary handwriting kinematic parameter (velocity) | Day 1
  Average absolute vertical velocity (cm/s)

SECONDARY OUTCOMES:
Secondary handwriting kinematic parameter (acceleration) | Day 1
  Average absolute vertical acceleration (cm/s²)
Secondary handwriting kinematic parameter (duration) | Day 1
  Average stroke duration (msec)
Pen pressure | Day 1
  Average pen pressure (levels)

CONTACTS AND LOCATIONS:
Locations (1):
- Aditya Murgai, London, Ontario, Canada